CLINICAL TRIAL: NCT06113341
Title: A Multi-centre, Prospective, Single-arm, Non-interventional Study Describing the Use of the Dose Check App in People Living With Type 2 Diabetes Mellitus and Treated With IDegLira in a Real-world Setting in Italy
Brief Title: A Research Study in Italy to Understand How the Dose Check App Used With Xultophy® Works in the Treatment of People Living With Type 2 Diabetes
Status: Withdrawn | Type: Observational
Why Stopped: The study has been cancelled due to the study's rejection from the local Italian ethics Committee
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-7589; U1111-1288-8131 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira; Xultophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IDegLira + Dose Check: Participants will be treated with commercially available Xultophy® (IDegLira) used with Dose Check app according to local label and routine clinical practice at the discretion of the treating physician.
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — Pre-filled pen injection.
  Other Names: Xultophy

SUMMARY:
This study will look at how a mobile based app called 'Dose Check' used along with Xultophy® helps the treatment in participants with type 2 diabetes mellitus (T2DM). Participants will get Xultophy® as prescribed by study doctor or will continue already prescribed treatment with Xultophy®. Participants will also be prescribed to use Dose Check app by study doctor. Participants will be asked to install the Dose Check app in their mobile phone, which will be supported with the correct dose of Xultophy®. The study will last for about 6 to 8 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 21 years at the time of signing informed consent.
* Diagnosed with T2DM >=12 weeks prior to signing consent.
* The decision to initiate treatment with commercially available Dose Check app as a part of treatment along with Xultophy® as per the local label has been made by the patient and the treating physician before and independently from the decision to include the participant in this study.
* Participants who are insulin naive (including the following situations: i. already on treatment with Xultophy® at V1 for less than or equal to (<=) 12 months and for <= 15 dose steps and ii. short-term insulin use for acute illness for a total of <14 days)
* Available HbA1c value <=12 weeks prior to the 'Informed consent and initiation of Dose Check app visit' (V1) or HbA1c measurement taken in relation with the 'Informed consent and initiation of Dose Check app visit' (V1), if in line with local clinical practice.
* Willingness to continue using the Dose Check app on a compatible smartphone according to the intended use for the entire duration of the study.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having signed informed consent in this study.
* Women known to be pregnant or breastfeeding, or women planning to become pregnant during the conduct of the study.
* Treatment with any investigational drug or software as a medical device (SaMD) within 30 days prior to enrolment into the study.
* Diagnosed with type 1 diabetes mellitus.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
* Hypersensitivity to the active substance or any of the excipients as specified in the Xultophy® local label.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants diagnosed with T2DM greater than or equal to (>=) 12 weeks and aged >=21 years at the time of signing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-11-07 (Estimated); Primary Completion 2025-02-23 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Participant downloaded and actively used the app (Yes/No) | From baseline (week 0) to end of the study (EOS) visit (week 26)
  Measured as count of participants.

SECONDARY OUTCOMES:
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to EOS visit (week 26)
  Measured as percentage (%) points.
Participants reaching individual HbA1c target set by physician | At EOS visit (week 26)
  Measured as count of participants (yes/no).
Participants reaching physician set individual fasting blood glucose (FBG) target | From baseline (week 0) to EOS visit (week 26)
  Measured as count of participants (yes/no).
Time to physician set individual FBG target from first reported FBG | From baseline (week 0) to EOS visit (week 26)
  Measured in number of weeks.
Participants achieving target level FBG according to clinical guidance | From baseline (week 0) to EOS visit (week 26)
  Measured as count of participants (yes/no).
Change in laboratory measured FPG | From baseline (week 0) to EOS visit (week 26)
  Measured in milligrams per deciliter (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (19):
- Italy (19):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro, Cz
  - Azienda Ospedaliero Universitario Policlinico "G. Martino", Gazi, ME
  - Azienda Ospedaliera Cannizzaro, Catania, Sicily
  - A.O. SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliera Ospedale Policlinico Consorziale, Bari
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - Ospedale di Chivasso, Chivasso
  - Presidio Ospedale di Cittadella Azienda ULSS 6 Euganea, Cittadella
  - Ospedale Santa Croce, Fano
  - Presidio Ospedaliero Santa Barbara, Iglesias
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
  - Ospedale San Francesco d'Assisi, Oliveto Citra
  - ARNAS Ospedali Civico Di Cristina Benfratelli, Palermo
  - Azienda Ospedaliero Universitaria Pisana Ospedale Cisanello, Pisa
  - Nuovo Ospedale degli Infermi, Ponderano
  - DIABETOLOGIA Ravenna AUSL della Romagna, Ravenna
  - AUSL Reggio Emilia, Reggio Emilia
  - A.O.U. Policlinico Umberto I, Roma
  - Fondazione Univ. Policlinico A.Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com